CLINICAL TRIAL: NCT00671554
Title: Phase II, Open-Label Trial in Patients With Stage IV Malignant Melanoma Using Melaxin as a Cancer Vaccine in Conjunction With BCG
Brief Title: Trial of Melaxin Cancer Vaccine Plus Bacillus Calmette-Guerin (BCG) to Treat Malignant Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to business considerations; not due to toxicities or adverse events.
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Oncolix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC/ORI 07-02
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma
Keywords: Melanoma; Dendritic cells; Cell therapy; BCG vaccine
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melaxin and BCG (Experimental): Four 1 ml doses of 250,000 dendritomas SQ at 4 week intervals along with a separate SQ injection containing 1 million Colony Forming Units (CFU) of BCG. The dose of BCG will be decreased by 50% in subsequent dosing if there is injection site ulceration
  Interventions: Biological: Melaxin (autologous dendritoma vaccine) and BCG

INTERVENTIONS:
Biological: Melaxin (autologous dendritoma vaccine) and BCG — Four 1 ml doses of 250,000 dendritomas SQ at 4 week intervals along with a separate SQ injection containing 1 million CFU of BCG. The dose of BCG will be decreased by 50% in subsequent dosing if there is injection site ulceration.
  Other Names: Melaxin

SUMMARY:
The purpose of this study is to determine if treatment with the autologous cellular vaccine, Melaxin, in combination with Bacillus Calmette-Guerin (BCG) injections is effective in Stage IV malignant melanoma.

DETAILED DESCRIPTION:
Chemotherapy and immunotherapy are the main therapies for metastatic melanoma with the hope of prolonging survival. The ideal immunotherapy would consist of the professional antigen-presenting cell, the dendritic cell, with the entire repertoire of tumor antigens inside. The best way to achieve this is by creating an autologous hybrid fusion cell of the dendritic cell and tumor cell. In this study, melanoma tumor tissue surgically removed from the patient will be disassociated into single cells, irradiated and fused to dendritic cells produced by culturing the patient's blood monocytes. Prior to the electrofusion procedure, the tumor cells are stained red and the dendritic cells are stained green. After fusion, the uniquely colored fused cells, or dendritomas, are separated from the unfused cells by use of a fluorescence activated cell sorter. This highly purified population is then divided into 4 doses containing 250,000 dendritomas each and frozen. Each dose is thawed, diluted to 1 milliliter (ml) with Sterile Saline for Injection containing 5 percent (%) human serum albumin and administered subcutaneously (SQ) over a lymph node bed to the patient once every 4 weeks. A separate injection of Bacillus Calmette-Guerin (BCG) is administered in the same area within 10 minutes of the dendritoma injection. The safety and efficacy of the therapy will be evaluated in 25 patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Male or female patient whose age is > 18 years of age
* Histological documented Stage IV malignant melanoma (American Joint Committee on Cancer (AJCC) sixth edition)
* Pathology report from tumor specimen verifying melanoma diagnosis
* Free of infection
* Hemoglobin> 9.0 grams per deciliter (gm/dL), White Blood Cells (WBC) >3000/ cubic millimeters (mm3), platelets> 100,000mm3
* Liver function test that are less than 2 times the upper limit of normal of the reference range for the testing laboratory
* Adequate cardiac function-any evidence of ischemic heart disease demonstrated by history, physical, or EKG will require referral to a cardiologist for evaluation and clearance prior to protocol therapy
* No immunotherapy within the past 3 months
* A minimum of 4 doses of lot-released, autologus Melaxin (1.0 million dendritomas)

Exclusion Criteria:

* Other malignancies in the past 5 years with the exception of non-melanoma skin cancer or carcinoma in situ of the cervix
* Has received any immunosuppressive agent within 30 days prior to treat
* Creatinine> 2.5 milligrams per deciliter (mg/dL) or currently on dialysis
* Positive serum pregnancy test, breast-feeding,or planning to conceive or father or father a child in the period surrounding the study as described in the informed consent.
* Women of childbearing potential who cannot follow the directions for birth control
* Eastern Cooperative Oncology Group (ECOG) performance status greater than 3
* Positive Rdonr panel (Human Immunodeficiency virus (HIV) 1, 2; Human T-lymphotropic virus (HTLV-1,2); Hepatitis B and C)
* History of a seizure disorder
* Brain metastases that have progressed within the last 6 months
* No measurable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Wagner, PhD, Study Director — Greenville Hospital System
Locations (1):
- Cancer Center of Carolinas/Clinical Research Unit 3rd Floor, Greenville, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Melaxin: Melaxin vaccine in conjunction with Bacillus Calmette-Guerin (BCG). Four 1 ml doses of 250,000 dendritomas Subcutaneous (SQ) at 4 week intervals along with a separate SQ injection containing 1 million Colony Forming Units (CFU) of BCG. The dose of BCG will be decreased by 50% in subsequent dosing if there is injection site ulceration.
Period: Overall Study
Arm/Group | Melaxin
Started | 3
Completed | 0
Not Completed | 3
Not completed — Disease progression | 3

BASELINE CHARACTERISTICS:
Groups:
- Melaxin: Melaxin vaccine in conjunction with Bacillus Calmette-Guerin (BCG)
Arm/Group | Melaxin
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (5.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Number of Participants With Unexpected Adverse Events or Unexpected Laboratory Results.
Description: Expected adverse events included injection site reactions, fever, chills, and arthralgias as anticipated with vaccine therapy. No unexpected or uncommon adverse events occurred such as disseminated sepsis. Clinical laboratory results on all participants were within expected ranges, including an increase in the number of IFN gamma expressing T-cells.
Time Frame: From first vaccine to 18 months after the last injection
Measure: Number; unit: participants
Arm/Group | Melaxin
Number analyzed (Participants) | 3
participants | 0

2. Secondary Outcome: Tumor Response Measured by RECIST Criteria and Progression-free Survival.
Description: CT scans for disease assessment occurred at three month intervals. If partial or complete responses were observed confirmation scans were performed within four weeks. Patients were followed for 18 months post study completion. All three participants recieved at least one vaccine, and all participants had progression of disease prior to the 18 month followup visit.
Time Frame: From first vaccine to 18 months after the last injection
Measure: Number; unit: participants
Arm/Group | Melaxin and BCG
Number analyzed (Participants) | 3
participants | 0

ADVERSE EVENTS:
Time Frame: first dose to 6 weeks after last dose
Arm/Group | Melaxin
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melaxin (N=3)
Brain Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Post-Operative meningitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Post-operative wound infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
injection site reactions (Skin and subcutaneous tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melaxin (N=3)
nausea (Gastrointestinal disorders) | 2 (2)
fatigue (General disorders) | 2 (2)
Injection site reactions (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No